CLINICAL TRIAL: NCT07286981
Title: Assessment of the Glycemic Index of Various Saudi Date Cultivars and Date-based Products. in Healthy Adults
Brief Title: Glycemic Index of Date Cultivars and Date-based Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Maha Alhussain, Associate Professor, King Saud University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 24/1428
Record Dates: First submitted 2025-12-03; First posted 2025-12-16 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-05

CONDITIONS: Glycaemic Response Measurements
Keywords: glycemic index; Glycemic load; Dates; Tamer; Rutab; Date paste; Date molasses

STUDY DESIGN:
Intervention Model Description: This is a randomized crossover interventional study, where each participant serves as his or her own control. All volunteers consume the reference glucose solution on three occasions and then consume each date product in separate sessions. After each test food, blood glucose is measured repeatedly over 120 minutes to determine the postprandial responses and subsequently calculate the glycemic index and glycemic load.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Group - Crossover Consumption of Date Products and Glucose Reference (Experimental): All participants will receive the glucose reference solution on three separate occasions and will consume the date or date-based product in individual sessions. Participants serve as their own control in a crossover design. Capillary blood glucose will be measured at several time points (0-120 minutes) after consumption to assess the glycemic index and load for each product.
  Interventions: Other: Date Cultivars and Date-based Products

INTERVENTIONS:
Other: Date Cultivars and Date-based Products — Participants will consume 50 g of available carbohydrates from each date or date-based product, including 13 Tamer varieties, 12 Rutab varieties, 3 types of date paste, and 3 types of date molasses. Each product will be tested in a separate session.. The intervention will also include consumption of a glucose reference solution (50 g glucose) on three separate occasions.
  Other Names: Tamer; Rutab; Date paste; Date molasses

SUMMARY:
Dates are widely consumed worldwide and hold substantial cultural importance in many Middle Eastern communities. Despite growing interest in measuring the glycemic response and glycemic index of foods for both research and practical applications, studies examining the glycemic properties of different date cultivars and their derived products remain limited. This study aims to determine the glycemic index (GI) and glycemic load (GL) of commonly consumed Saudi date cultivars and their derived products in healthy subjects, and to evaluate their potential impact on postprandial glucose responses. The study will consist of 4 phases as follows: phase 1: Date varieties at Tamer stage; phase 2: date varieties at Rutab stage; phase 3: Date's debs; phase 4: Date's paste. For each phase, ten subjects will be asked to attend the laboratory in the morning after an overnight fast on several occasions. Each visit will be separated from the next by a "washout" day. The reference food, 50 g of glucose dissolve in 250 ml water will be tested on 3 alternating days to diminish day to day variation of glucose tolerance. 50g equivalent carbohydrates of dates will be consumed with 250 ml of water. Participants will be blinded to the type of the dates. Glucose will be measured in capillary blood samples following the two hours of the test meal consumption, at 15 min interval (0, 15, 30, 45, 60, 90 and 120 min) . A qualified technician will perform all blood glucose measurements.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 to 55 years
* Normotensive (normal blood pressure)
* Normal fasting glucose levels
* Not taking any prescription medication
* Able and willing to provide written informed consent

Exclusion Criteria:

* Morbid obesity (BMI > 40 kg/m²)
* Pre-diabetic status
* Pregnancy
* Any gastrointestinal disorders
* History of gastroenteritis within the preceding six months
* Previous gastrointestinal surgeries
* Smoking
* Presence of chronic conditions (e.g., asthma, rheumatoid arthritis)
* Presence of acute illnesses (e.g., respiratory or urinary tract infections)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-08-16 (Actual); Primary Completion 2025-05-25 (Actual); Study Completion 2025-05-25 (Actual)

PRIMARY OUTCOMES:
Glycemic Index | Baseline (fasting) and up to 120 minutes post-consumption on each test day.
  The glycemic index of each date cultivar and date-based product will be determined on designated test days by calculating the incremental area under the blood glucose response curve (iAUC) over the 120-minute postprandial period following consumption of a portion containing 50 g of available carbohydrates, relative to the iAUC of a reference glucose solution. Blood glucose measurements will be obtained at baseline (fasting) and at predefined time points up to 120 minutes after ingestion.

SECONDARY OUTCOMES:
Glycemic Load (GL) of Fresh and Processed Date Products | Baseline (fasting) and up to 120 minutes post-consumption on each test day.
  The glycemic load of each date-based product will be calculated on each test day using the measured glycemic index and the available carbohydrate content of a typical serving, based on blood glucose measurements obtained at baseline and up to 120 minutes post-consumption.

CONTACTS AND LOCATIONS:
Overall Officials: Maha Alhussain, PhD, Study Director — King Saud University
Locations (1):
- King Saud University, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
Notably, individual participant data will not be shared to ensure the privacy and confidentiality of the study participants. The data includes personal health information and making them publicly available might risk the identification of participants despite efforts to anonymize them.

REFERENCES:
- [Background] Brouns F, Bjorck I, Frayn KN, Gibbs AL, Lang V, Slama G, Wolever TM. Glycaemic index methodology. Nutr Res Rev. 2005 Jun;18(1):145-71. doi: 10.1079/NRR2005100. PMID 19079901